CLINICAL TRIAL: NCT06677606
Title: The Analgesic Efficacy of Pericapsular Nerve Group Block (PENG) in Comparison With Periarticular Local Anesthetic Infiltration (PAI) Undergoing Hip Hemiarthroplasty : a Randomized Controlled Study
Brief Title: PENG Block in Comparison With Anesthetic Infiltration (PAI) After Hip Hemiarthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Yasser S Mostafa, MD, Lecturer of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D370
Record Dates: First submitted 2024-11-02; First posted 2024-11-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain
Keywords: PENG bock; PAI block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block group (Experimental): patients will receive PENG block after skin closure, .Patients will be placed in the supine position. The ultra sound transducer will be placed in a transverse orientation, medial and caudal to the anterosuperior iliac spine in order to identify the anteroinferior iliac spine, the iliopubic eminence and the psoas tendon. Using an in-plane technique and a lateral-to-medial direction, the block needle will be advanced until its tip will be positioned on the periosteum dorsal to the psoas tendon. The LA (20mL of bupivacaine 0.5%) will be injected following negative aspiration.. The accurate position of the needle was confirmed by hydro dissection and spread under the illo-psoas muscle .
  Interventions: Procedure: PENG block
- PAI group (Active Comparator): PIA BLOCK For subjects randomized to PAI , LA infiltration will be carried out using a total dose of 150mg of bupivacaine and a total volume of 60mL. The admixture (consisting of 60mL of bupivacaine 0.25% and 30mg of ketorolac) will be loaded into two 30mL syringes at the beginning of surgery. After insertion of the acetabular component (and before insertion of the femoral stem), the surgeon will infiltrate the deep tissues (ie, anterior and posterior capsules, gluteus minimus and medius muscles, supraacetabular region, area around the anterior inferior iliac spine, and quadratus femoris muscle all the while avoiding the deep hip external rotator muscle group in order to prevent sciatic nerve block) with the first 30mL syringe. Before wound closure, the gluteus maximus muscle, iliotibial band, subcutaneous tissues, and skin will be infiltrated with the second 30mL syringe.
  Interventions: Procedure: PAI block

INTERVENTIONS:
Procedure: PENG block — The ultra sound transducer will be placed in a transverse orientation, medial and caudal to the anterosuperior iliac spine in order to identify the anteroinferior iliac spine, the iliopubic eminence and the psoas tendon. Using an in-plane technique and a lateral-to-medial direction, the block needle will be advanced until its tip will be positioned on the periosteum dorsal to the psoas tendon. The LA (20mL of bupivacaine 0.5%) will be injected following negative aspiration.. The accurate position of the needle was confirmed by hydro dissection and spread under the illo-psoas muscle
  Arms: PENG block group
Procedure: PAI block — LA infiltration will be carried out using a total dose of 150mg of bupivacaine and a total volume of 60mL. The admixture (consisting of 60mL of bupivacaine 0.25% and 30mg of ketorolac) will be loaded into two 30mL syringes at the beginning of surgery. After insertion of the acetabular component (and before insertion of the femoral stem), the surgeon will infiltrate the deep tissues (ie, anterior and posterior capsules, gluteus minimus and medius muscles, supraacetabular region, area around the anterior inferior iliac spine, and quadratus femoris muscle all the while avoiding the deep hip external rotator muscle group in order to prevent sciatic nerve block) with the first 30mL syringe. Before wound closure, the gluteus maximus muscle, iliotibial band, subcutaneous tissues, and skin will be infiltrated with the second 30mL syringe.
  Arms: PAI group

SUMMARY:
The goal of this intervention study is to compare the analgesic efficacy of pericapsular nerve group (PENG) block versus periarticular anesthetic infiltration (PAI) block in patients undergo hemiarthroplasty after spinal anesthesia .

The main questions it aims to answer are:

which block has more analgesic efficacy. which block has more motor-sparing analgesia.

Researchers will compare optimal motor-sparing analgesia between PENG block and PAI after hemiarthroplasty.

Participants will be divided in two groups :

group receive PENG block and other group receive PAI

DETAILED DESCRIPTION:
This study aims to compare the analgesic efficacy of pericapsular nerve group (PENG) block versus periarticular anesthetic infiltration (PAI) block in hemiarthroplasty after spinal anesthesia

PARTICIPANTS AND METHODS:

After approval of the local institutional ethics committee and local institutional review board. Patients who are scheduled for elective hemiarthroplasty and fulfilling the inclusion criteria in Fayoum university hospital starting from October 2024 will be enrolled in this randomized controlled study until fulfilling sample size. A detailed informed consent will be signed by the eligible participants before recruitment.

Inclusion criteria The eligibility criteria included ages from 50 to 90 years, American Society of Anesthesiologists (ASA) physical status I to III, and undergoing bipolar hemiarthroplasty in Fayoum university hospital.

Exclusion criteria Patient refusal, contraindication to spinal anesthesia , clinically significant coagulopathy, infection at the injection site, allergy to local anesthetics, body mass index>35 kg m2 , diabetic or other neuropathies, patients receiving opioids for chronic analgesic therapy

. ANESTHETIC TECHNIQUE Perioperative anesthesia management will be according to our hospital routine protocol. An intravenous cannula will be inserted in the hand and standard monitoring (noninvasive blood pressure, electrocardiography, and pulse oximetry) will be applied . In all patients, spinal anesthesia will be performed in the sitting position. The midline and level of the L3-4 and L4-5 intervertebral spaces will be identified, and spinal anesthesia will be administered using 10 mg of isobaric bupivacaine (2mL of bupivacaine 0.5%) injected using 25-gauge Quincke needle. Patients will be immediately placed in the supine position. Spinal anesthesia will be considered successful when a bilateral block to T12, as assessed by loss of cold (cold ice) and pain (a 23-gauge needle) sensations, will be established 10 minutes after the intrathecal injection., the bipolar hemiarthroplasty will be performed in all patients in nondependent lateral position.

Randomization and blinding Using a computer-generated sequence of random numbers and a sealed, opaque envelope technique, patients will be randomly allocated to receive PENG block or PAI . The randomization list and opaque envelopes will be created by an assistant who will not be involved in patient care.

Performance of PENG blocks and PAI PENG BLOCK will be performed in the operating room, after skin closure, .Patients will be placed in the supine position. The ultra sound transducer will be placed in a transverse orientation, medial and caudal to the anterosuperior iliac spine in order to identify the anteroinferior iliac spine, the iliopubic eminence and the psoas tendon. Using an in-plane technique and a lateral-to-medial direction, the block needle will be advanced until its tip will be positioned on the periosteum dorsal to the psoas tendon. The LA (20mL of bupivacaine 0.5%) will be injected following negative aspiration.. The accurate position of the needle was confirmed by hydro dissection and spread under the illo-psoas muscle .

PIA BLOCK For subjects randomized to PAI , LA infiltration will be carried out using a total dose of 150mg of bupivacaine and a total volume of 60mL. The admixture (consisting of 60mL of bupivacaine 0.25% ) will be loaded into two 30mL syringes at the beginning of surgery. After insertion of the acetabular component (and before insertion of the femoral stem), the surgeon will infiltrate the deep tissues ( anterior and posterior capsules, gluteus minims and Medius muscles, supraacetabular region, area around the anterior inferior iliac spine, and quadratus fumoirs muscle all the while avoiding the deep hip external rotator muscle group in order to prevent sciatic nerve block) with the first 30mL syringe. Before wound closure, the gluteus maximus muscle, iliotibial band, subcutaneous tissues, and skin will be infiltrated with the second 30mL syringe

Statistical analysis and sample size estimation Before conducting the study, G*Power 3.1.9.6 will be utilized to establish the appropriate sample size for equal distribution among the two groups based on data from the study by Bravo et al. who recorded median and range between the same two groups for numeric rating scale at 12 hours which is our primary outcome. We convert and calculate these numbers to mean from Luo et al. (2018) and standard deviation from Wan et al. (2014) and found a mean difference of 1.75 and standard deviation of 2.45 and 1.97 for the two study groups creating effect size of 0.78. Depending on a significance level (α) of 0.05, a power (1 - β) of 0.80, allocation ratio 1:1 and two-tailed, a sample size of 27 patients is required for each group. Due to the possibility of dropout rate and exclusion of some objects, the study will be planned to include 60 patients (30 patients in each group).

Statistical analysis will be conducted using IBM SPSS Statistics 22 (IBM Corp., Armonk, NY, USA). The normal distribution of data will be assessed by the Kolmogorov-Smirnov and Shapiro-Wilk tests. Mean and standard deviation will be used as descriptive statistics for normally distributed numerical variables, while median and interquartile range (25th to 75th percentiles) will be used as descriptive statistics for non-normally distributed numerical variables. In addition, Chi-square test will be employed to test the significance between categorical variables. Independent t test will be employed for numerical data that exhibited normal distribution, whereas the Mann Whitney test will be used for numerical data that did not adhere to normal distribution. A significance level of p < 0.05 will be deemed to be statistically significant

ELIGIBILITY:
Inclusion Criteria:

ages from 50 to 90 years and undergoing bipolar hemiarthroplasty in Fayoum university hospital American Society of Anesthesiologists (ASA) physical status I to III,.

Exclusion Criteria:

Patient refusal. contraindication to spinal anesthesia . clinically significant coagulopathy. infection at the injection site. allergy to local anesthetics. body mass index>35 kg m2., diabetic or other neuropathies. patients receiving opioids for chronic analgesic therapy.

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
the pain score (NRS) | at 12 hours after injection of local anethesia
  the pain score (NRS) after surgery at rest (score 0 =no pain and 10 =worst pain ever) .

SECONDARY OUTCOMES:
the pain score (NRS) | at 6, 18, 24, and 48 hours after injection of local anethesia
  the pain score (NRS) after surgery at rest (score 0 =no pain and 10 =worst pain ever)
Incidence of quadriceps motor block | at 3,6,24 hours after injection of local anesthesia
  paresis or paralysis of knee extension) at 3,6,24 hours postoperatively. Knee extension Will be evaluated in a supine position with the patient's hip and knee flexed at 45° and 90°, respectively. The patient will be asked to extend the knee first against gravity and then against resistance. Knee extension will be graded according to a 3-point scale: 0=normal strength (extension against gravity and against resistance); 1=paresis (extension against gravity but not against resistance); 2=paralysis (no extension possible
cumulative morphine consumption in 24 hours. | at 24 hours after injection of local anethesia
  net total doses of morphine used after surgery
The incidence of block-related adverse events (ie, vascular puncture, LA toxicity). | at 24 hours after injection of local anethesia
  complication of injection of local anethesia (ie, vascular puncture, toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Natrajan P, Bhat RR, Remadevi R, Joseph IR, Vijayalakshmi S, Paulose TD. Comparative Study to Evaluate the Effect of Ultrasound-Guided Pericapsular Nerve Group Block Versus Fascia Iliaca Compartment Block on the Postoperative Analgesic Effect in Patients Undergoing Surgeries for Hip Fracture under Spinal Anesthesia. Anesth Essays Res. 2021 Jul-Sep;15(3):285-289. doi: 10.4103/aer.aer_122_21. Epub 2022 Feb 7. PMID 35320956
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Senthil KS, Kumar P, Ramakrishnan L. Comparison of Pericapsular Nerve Group Block versus Fascia Iliaca Compartment Block as Postoperative Pain Management in Hip Fracture Surgeries. Anesth Essays Res. 2021 Oct-Dec;15(4):352-356. doi: 10.4103/aer.aer_119_21. Epub 2022 Mar 1. PMID 35422548
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Bravo D, Aliste J, Layera S, Fernandez D, Erpel H, Aguilera G, Arancibia H, Barrientos C, Wulf R, Leon S, Branes J, Finlayson RJ, Tran Q. Randomized clinical trial comparing pericapsular nerve group (PENG) block and periarticular local anesthetic infiltration for total hip arthroplasty. Reg Anesth Pain Med. 2023 Oct;48(10):489-494. doi: 10.1136/rapm-2023-104332. Epub 2023 Feb 16. PMID 36797036
- [Background] Ye S, Wang L, Wang Q, Li Q, Alqwbani M, Kang P. Comparison between Ultrasound-Guided Pericapsular Nerve Group Block and Local Infiltration Analgesia for Postoperative Analgesia after Total Hip Arthroplasty: A Prospective Randomized Controlled Trial. Orthop Surg. 2023 Jul;15(7):1839-1846. doi: 10.1111/os.13777. Epub 2023 Jun 29. PMID 37382431
- [Background] Hu J, Wang Q, Hu J, Kang P, Yang J. Efficacy of Ultrasound-Guided Pericapsular Nerve Group (PENG) Block Combined With Local Infiltration Analgesia on Postoperative Pain After Total Hip Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2023 Jun;38(6):1096-1103. doi: 10.1016/j.arth.2022.12.023. Epub 2022 Dec 16. PMID 36529195